CLINICAL TRIAL: NCT06553456
Title: Random, Double-blind, Parallel Group Phase II/III Clinical Trial to Evaluate the Effectiveness and Safety of Recombinant Human Serum Albumin Versus Human Serum Albumin in Hepatic Cirrhosis Patients With Ascites
Brief Title: Phase II/III Clinical Trial of Recombinant Human Serum Albumin in Cirrhotic Patients With Ascites
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Protgen Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: rHSA 2020-3 (Phase Ⅲ)
Record Dates: First submitted 2024-08-11; First posted 2024-08-14 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-09

CONDITIONS: Cirrhotic Ascites
MeSH Terms: interventions — recombinant human serum albumin-heme; Serum Albumin, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): The experimental drug was administered at a dose of 20 g/ day for 7 days.
  Interventions: Drug: Recombinant Human Serum Albumin
- Group 2 (Active Comparator): The positive control drug was administered at a dose of 20 g/ day for 7 days.
  Interventions: Drug: Human Serum Albumin

INTERVENTIONS:
Drug: Recombinant Human Serum Albumin — The experimental drug was administered at a dose of 20 g/ day for 7 days.
  Arms: Group 1
Drug: Human Serum Albumin — The positive control drug was administered at a dose of 20 g/ day for 7 days.
  Arms: Group 2

SUMMARY:
This trial adopts random, double-blind, positive control, parallel group design to evaluate the effectiveness and safety of recombinant human serum albumin versus human serum albumin in hepatic cirrhosis patients with ascites.

DETAILED DESCRIPTION:
This trial adopts random, double-blind, positive control, parallel group design to evaluate the effectiveness and safety of recombinant human serum albumin versus human serum albumin in hepatic cirrhosis patients with ascites.

In this trial（phase III）, the efficacy of rHSA will be evaluated by the change in serum albumin concentration immediately after the last intravenous administration from baseline, and its safety, PD characteristics and immunogenicity will be further evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Agree to follow the experimental treatment plan and visit schedule, voluntarily join the group, and sign a written informed consent form;
2. On the day of signing the informed consent form, the age is between 18 and 70 years old, and there is no gender limit; Body mass index (BMI) within the range of 17.0-29.0 kg/m² (including boundary values);
3. Patients diagnosed clinically with decompensated liver cirrhosis ascites, and confirmed by abdominal ultrasound examination during screening to have ascites grading of 1-2, while meeting the requirement of serum albumin (ALB)<30 g/L;
4. Men with fertility and women of childbearing age (women of childbearing age include premenopausal women and women within two years after menopause) are willing to take effective contraceptive measures (condoms, contraceptive sponges, contraceptive gel, contraceptive membranes, intrauterine devices, oral or injectable contraceptives, subcutaneous implants, etc.) within three months after the last administration of the trial drug from the date of signing the informed consent; Women of childbearing age must have a negative pregnancy test result within ≤ 7 days before the first trial drug administration.

Exclusion Criteria:

1. Individuals with a known history of allergies/allergic reactions to yeast or yeast derived products, or those who are allergic to any component of the study formulation; Individuals with an allergic constitution (multiple drug or food allergies) or a history of allergies to biological products, as well as a history of severe systemic allergic reactions caused by other reasons and deemed unsuitable for treatment with the investigational drug by the researcher;
2. During the screening process, there were serious digestive system diseases and complications that the researchers deemed unsuitable for participation in this study, including but not limited to malignant ascites, diagnosis of grade III or IV hepatic encephalopathy according to the West Haven grading criteria, portal vein cancer thrombus/thrombus, circulatory dysfunction after abdominal puncture, biliary obstructive disease determined by ultrasound or other imaging examinations, gastrointestinal bleeding that stopped bleeding after treatment for less than 10 days or endoscopic ligation could not effectively stop bleeding, or those assessed by the researchers as having a high risk of bleeding during the trial period (such as severe esophagogastric varices with positive red sign on gastroscopy within 3 months before screening);
3. When screening, there is a history of active cardiovascular disease or other conditions that researchers determine are not suitable for receiving human serum albumin treatment, including but not limited to hypertension (systolic blood pressure>140 mmHg or diastolic blood pressure>90 mmHg, except for those determined by researchers to have good medication control and stable condition), severe anemia, acute heart disease, severe cardiovascular or structural heart disease, severe arrhythmia, decompensated heart failure (normal blood volume or high blood volume), unstable angina pectoris, myocardial infarction in the past 6 months before screening, tachycardia/bradycardia requiring medication treatment, third degree atrioventricular block, etc;
4. Active metabolic system disease or medical history (except for diabetes patients with stable blood glucose control as judged by the investigator), or combined with renal function injury, which is not suitable for serum albumin treatment as judged by the investigator;
5. When screening, there were serious underlying diseases that the researchers deemed unsuitable for participation in this study, including but not limited to active malignant tumors (including hepatocellular carcinoma [HCC]), pulmonary edema, bleeding tendency or active bleeding disease, uncontrolled infections (including active spontaneous bacterial peritonitis [SBP1]), thyroid dysfunction (according to the National Cancer Institute's Common Terminology Criteria for Adverse Events INCICTCAEI 5.0 grade 3 or above), pleural effusion that the researchers determined may require treatment or have disease changes throughout the entire trial process, etc;
6. The patient has the following laboratory test abnormalities: (1) Bone marrow function: Absolute neutrophil count (ANC)<1.0x10 ^ 9/L; Platelets (PLT)<20x10 ^ 9/L; Hemoglobin (HGB)<70gL; (2) Liver function: Alanine aminotransferase (ALT)>5 × ULN (upper limit of normal); Aspartate aminotransferase (AST)>5 × ULN; Serum bilirubin (TBIL)>4 x upper limit of normal (ULN) or deemed unsuitable for participation in the trial by the researcher; (3) Renal function: serum creatinine>3 times the upper limit of normal (ULN), positive urine protein, and the researcher's judgment that it is not suitable to participate in the trial; (4) Coagulation function: prothrombin time (PT) prolonged>5s；
7. Individuals who have received human plasma preparations (including human albumin preparations) within 7 days prior to the first administration of the investigational drug; Individuals with a history of organ transplantation; Those who need to undergo or plan invasive invasive examinations or treatments during the research period;
8. Participated in or was participating in clinical trials of other new drugs or medical devices within 30 days prior to screening, and used the investigational drug/treatment provider;
9. Individuals who test positive for human immunodeficiency virus (HIV) antibodies;
10. Pregnant or lactating women;
11. Other reasons why researchers believe it is not suitable to participate in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Actual)
Dates: Start 2024-08-19 (Actual); Primary Completion 2025-05-14 (Actual); Study Completion 2025-05-14 (Actual)

PRIMARY OUTCOMES:
Change of serum albumin concentration | 7 days
  The change in serum albumin concentration confirmed by albumin examination immediately after the completion of secondary intravenous administration compared to baseline (based on the results of central laboratory tests)

SECONDARY OUTCOMES:
Key Secondary Outcome Measures: The improvement rate of ascites | 7 days
  The improvement rate of ascites at the completion of the last intravenous administration
The change in serum albumin concentration immediately after completion of the last intravenous dose, as confirmed by albumin testing at the local laboratory | 7 days
  The change in serum albumin concentration confirmed by local laboratory albumin test immediately after the last intravenous administration compared to baseline
Changes in the depth of ascites | 7 days
  Changes in ascites depth from baseline upon completion of the last intravenous administration
The proportion of subjects with serum albumin concentration ≥ 35 g/L | 7 days
  The proportion of subjects whose serum albumin concentration confirmed by albumin examination at the completion of the last intravenous administration is ≥ 35 g/L
The time when serum albumin concentration reached ≥35 g/L | 90 days
  The time when serum albumin concentration reached ≥35 g/L
Changes in abdominal circumference | 7 days
  Changes in abdominal circumference compared to baseline at the completion of the last intravenous administration
Changes in body weight | 7 days
  Changes in body weight compared to baseline at the completion of the last intravenous administration
The change in serum albumin concentration during the re-treatment period | 7 days
  The change in serum albumin concentration confirmed by albumin examination immediately after the completion of the last intravenous administration during the re-treatment period compared to the baseline before the re-treatment
The improvement rate of ascites during the re-treatment period | 7 days
  The improvement rate of ascites at the completion of the last intravenous administration during the re-treatment period
Changes in the depth of ascites during the re-treatment period | 7 days
  Changes in ascites depth at the completion of the last intravenous administration during the re-treatment period compared to baseline before the re-treatment
The proportion of subjects with serum albumin concentration ≥ 35 g/L during the re-treatment period | 7 days
  Proportion of subjects with serum albumin concentration ≥ 35 g/L confirmed by albumin examination during the re-treatment period
The time when serum albumin concentration reached ≥35 g/L during the re-treatment period | 7 days
  The time when the serum albumin concentration confirmed by the albumin test during the re-treatment period reaches ≥ 35 g/L
Changes in abdominal circumference during the re-treatment period | 7 days
  Changes in abdominal circumference at the completion of the last intravenous administration during the re-treatment period compared to baseline before the re-treatment
Changes in body weight during the re-treatment period | 7 days
  Changes in body weight at the completion of the last intravenous administration during the re-treatment period compared to baseline before the re-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jidong Jia, Ph.D, Study Director — Beijing Friendship Hospital
Locations (1):
- Shenzhen Protgen Ltd, Guangdong, Shenzhen, China

IPD SHARING:
Plan to Share IPD: No